CLINICAL TRIAL: NCT04902521
Title: Concurrent Use of Transcranial Magnetic Stimulation and Constraint Induced Movement Therapy in Children With Unilateral Cerebral Palsy: A Feasibility Study
Brief Title: Use of Transcranial Magnetic Stimulation and Constraint Induced Movement Therapy in Pediatric Unilateral Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, M. Florencia Ricci, Principle Investigator, Developmental Pediatrician, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS24766(B2021:023)
Record Dates: First submitted 2021-04-22; First posted 2021-05-26 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; constrain induced muscle therapy; Transcranial magnetic stimulation
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcranial magnetic stimulation with constraint induced movement therapy (Experimental): CIMT/TMS: Five participants will receive a one-hour weekly occupational therapy session of CIMT with 2-hours of daily home program for a total of 6 weeks; immediately prior to initiation of each CIMT session, participants will receive 20 minutes of TMS 1HZ.
  Interventions: Device: Transcranial magnetic stimulation
- constraint induced movement therapy Sham transcrianial magnetic stimulation (Sham Comparator): (CIMT/sham TMS): Five participants will receive a one-hour weekly session of CIMT with 2-hours daily of home program for a total of 6 weeks; immediately prior to initiation of each CIMT session, participants will receive 20 minutes of sham TMS 1HZ.
  Interventions: Device: Sham Transcranial Magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (TMS) is a safe non-invasive technique that stimulates the brain using repetitive magnetic pulses to enhance neuroplasticity. TMS has been shown to produce lasting modulation of cortical activity and improve clinical symptoms of children with neurodevelopmental disorders including CP
  Other Names: TMS
  Arms: Transcranial magnetic stimulation with constraint induced movement therapy
Device: Sham Transcranial Magnetic stimulation — Sham Transcranial Magnetic stimulation will be given to the control group. During the Sham procedure patients will sit near the TMS but will not receive any magnetic pulses.
  Other Names: Sham TMS
  Arms: constraint induced movement therapy Sham transcrianial magnetic stimulation

SUMMARY:
Cerebral Palsy (CP) is the most common cause of childhood physical disability. Early CP diagnosis and intervention are crucial to improving outcomes in these patients. Constraint-induced movement therapy (CIMT) has become a standard therapeutic intervention for children with unilateral CP. CIMT utilizes restraining of the unaffected upper limb to stimulate the use of the paretic upper limb enhancing neuroplasticity in the affected cerebral hemisphere.

Transcranial magnetic stimulation (TMS) is a safe non-invasive technique that stimulates the brain using repetitive magnetic pulses to enhance neuroplasticity. TMS has been shown to improve symptoms of children with neurodevelopmental disorders such as CP. It is predicted that a combined therapy that uses CIMT and TMS is could improve mobility in children with unilateral CP.

To determine if combined therapy is beneficial to children with CP and if use of this therapy is feasible for families, the investigators would like to conducted a feasibility trial. In this trial the investigators will enrol 10 children who have unilateral CP, the participants will either receive:

1. CIMT and TMS or;
2. CIMT and fake TMS, fake TMS consist of a child sitting near the TMS machine but not receiving any TMS.

The aim of this project is to determine if it is feasible to conduct a large randomized control trial to compare the effects of combined CIMT and TMS versus CIMT and fake TMS.The investigators also hope that by conducting this trial they can identify any benefits that the addition of TMS may have in children with CP.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common cause of childhood physical disability. Early CP diagnosis and intervention are crucial in optimizing neuroplasticity and improving outcomes. One such intervention is constraint-induced movement therapy (CIMT), a therapeutic approach used in children with unilateral CP. CIMT utilizes restraining of the unaffected upper limb to stimulate the use of the paretic upper limb enhancing neuroplasticity in the affected cerebral hemisphere.CIMT is more effective than other rehabilitation approaches in improving upper limb function and has become a standard therapeutic intervention for children with unilateral CP.

Repetitive transcranial magnetic stimulation (TMS) is a safe non-invasive technique that stimulates the brain using repetitive magnetic pulses to enhance neuroplasticity. TMS has been shown to produce lasting modulation of cortical activity and improve clinical symptoms of children with neurodevelopmental disorders including CP.

A recent Canadian study, the PLASTIC Champs trial, demonstrated that combining TMS and CIMT for children with unilateral CP secondary to perinatal stroke produced greater improvements in upper limb function when compared to CIMT or TMS alone. Though promising, there are three features of the Plastic Champs trial that could limit its generalizability. First, it took place in a very special, intensive setting of daily CIMT/TMS during a 14-day camp. Second is the single cause of CP studied. And finally, it included only school-age children. To date, no research study has evaluated if findings from the PLASTIC Champs trial could be replicated when utilizing the combination of CIMT and TMS in a regular clinical environment, and among younger children.

A feasibility study is an appropriate first step towards our plan of performing a definitive RCT on the topic.

In this trial the investigators will enrol 10 children who have unilateral CP, they will either receive:

1. CIMT and TMS or;
2. CIMT and fake TMS, fake TMS consist of a child sitting near the TMS machine but not receiving any TMS.

The Investigators seek to evaluate whether, in younger children, the addition of TMS to the more commonly used, intermittent outpatient regimen of CIMT improves the motor outcomes of the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of unilateral spastic CP
* assessed as Gross Motor Function Classification System level I to III
* assessed as Manual Ability Classification System level II to level IV

Exclusion Criteria:

* have received CIMT in the last 6 month
* do not have neuroimaging studies to confirm clinical diagnosis of CP
* severe impairments limiting their ability to participate

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Participant recruitment | 5 Months
  Participant recruitment: We will assess number of eligible children, reasons for ineligibility and non-participation.
Evaluation of Participant retention during trial | 5 Months
  We will assess and report the number of missing variables and number of patients with incomplete outcome measures.
Incidence of Treatment-Emergent Adverse Events as assessed by Parental Reports | 5 Months
  We will ask parents to report weekly on the presence of previously reported side effects including headaches, anxiety, dizziness, tingling, mood changes, difficulties with concentration, abnormal muscle contractions, nausea, stomach ache, fatigue and decreased hand function of either hand. For completeness we will also ask about presence of seizures (new onset or increase in existing seizures), although this side effect was not seen in previous safety studies. We will also assess number of times (and reasons) TMS session ended before the stipulated time and number of minutes lost.
Effectiveness of the transcrainial magnetic stimulation blinding process on patients and therapist | 5 months
  TMS sham process and blinding of patients and therapist: At the end of the study we will ask parents/ occupational therapist assessing outcomes to report on possible group allocation of participant (could they identify if the participant received TMS or sham TMS?)
Evaluation of treatment intervention by parental guardians | 3 months
  Acceptability of treatment: Based on Gillick's work, at the end of the intervention (6 weeks) and 3 months post completion, we will ask parents to rate on a scale of 1 to 10 their "satisfaction with the intervention, willingness to repeat the study, and likelihood of recommending the study to others." .
  - Participant research engagement: At the end of the study we will ask parents to rate their willingness to participate as a research-collaborator in a future large RCT study.
Estimation of intervention costs | 5 months
  This study will provide information needed to develop a budget for the future application.

SECONDARY OUTCOMES:
Assessment of mobility using Small Kids-AHA | 5 months
  We will assess differences between pre-to post intervention using the Small Kids- AHA scores among those undergoing CIMT+TMS vs. CIMT/sham TMS. Small Kids-AHA is a measure of bimanual performance and is rated on a scale or 0-100 (100 being high functionality).
Assessment of mobility using the Canadian Occupational Performance Measure (COPM) | 5 months
  We will assess differences between pre-to post intervention using the Canadian Occupational Performance Measure (COPM) scores among those undergoing CIMT+TMS vs. CIMT/sham TMS. Canadian Occupational Performance Measure is used to asses daily functioning and is scored on a 10 point scale (10 being high functionality).

CONTACTS AND LOCATIONS:
Locations (1):
- SSCY/RCC, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Background] Gordon AM. To constrain or not to constrain, and other stories of intensive upper extremity training for children with unilateral cerebral palsy. Dev Med Child Neurol. 2011 Sep;53 Suppl 4:56-61. doi: 10.1111/j.1469-8749.2011.04066.x. PMID 21950396
- [Background] Uswatte G, Taub E. Constraint-induced movement therapy: a method for harnessing neuroplasticity to treat motor disorders. Prog Brain Res. 2013;207:379-401. doi: 10.1016/B978-0-444-63327-9.00015-1. PMID 24309263
- [Background] Chen YP, Pope S, Tyler D, Warren GL. Effectiveness of constraint-induced movement therapy on upper-extremity function in children with cerebral palsy: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2014 Oct;28(10):939-53. doi: 10.1177/0269215514544982. Epub 2014 Aug 14. PMID 25125440
- [Background] Sakzewski L, Ziviani J, Boyd RN. Efficacy of upper limb therapies for unilateral cerebral palsy: a meta-analysis. Pediatrics. 2014 Jan;133(1):e175-204. doi: 10.1542/peds.2013-0675. Epub 2013 Dec 23. PMID 24366991
- [Background] Eliasson AC, Holmefur M. The influence of early modified constraint-induced movement therapy training on the longitudinal development of hand function in children with unilateral cerebral palsy. Dev Med Child Neurol. 2015 Jan;57(1):89-94. doi: 10.1111/dmcn.12589. Epub 2014 Sep 19. PMID 25236758
- [Background] Masuda F, Nakajima S, Miyazaki T, Tarumi R, Ogyu K, Wada M, Tsugawa S, Croarkin PE, Mimura M, Noda Y. Clinical effectiveness of repetitive transcranial magnetic stimulation treatment in children and adolescents with neurodevelopmental disorders: A systematic review. Autism. 2019 Oct;23(7):1614-1629. doi: 10.1177/1362361318822502. Epub 2019 Jan 20. PMID 30663323
- [Background] Kirton A, Andersen J, Herrero M, Nettel-Aguirre A, Carsolio L, Damji O, Keess J, Mineyko A, Hodge J, Hill MD. Brain stimulation and constraint for perinatal stroke hemiparesis: The PLASTIC CHAMPS Trial. Neurology. 2016 May 3;86(18):1659-67. doi: 10.1212/WNL.0000000000002646. Epub 2016 Mar 30. PMID 27029628